CLINICAL TRIAL: NCT00080860
Title: Efficacy Of Sentinel Lymph Node Biopsy And Primary Tumor Gene Expression Profiling To Detect Axillary Lymph Node Metastases After Neoadjuvant Chemotherapy For Breast Cancer
Brief Title: Sentinel Lymph Node Biopsy and Primary Tumor Gene Expression Profiling in Finding Axillary Lymph Node Metastases in Women Who Have Received Neoadjuvant Therapy for Stage II, Stage III, or Stage IV Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 040114; 04-C-0114; CDR0000356050; NCT00076895 (obsolete NCT alias)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis; Immunohistochemistry; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

INTERVENTIONS:
Genetic: microarray analysis
Other: immunohistochemistry staining method
Procedure: conventional surgery
Procedure: lymphangiography
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: Sentinel lymph node biopsy and gene expression profiling of the primary breast tumor may help determine if tumor cells have spread to the axillary lymph nodes and help doctors plan more effective surgery for breast cancer.

PURPOSE: This clinical trial is studying how well sentinel lymph node biopsy and primary tumor gene expression profiling work in finding lymph node metastases in women who have received neoadjuvant therapy for stage II, stage III, or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sentinel lymph node mapping for assessing axillary lymph node status after neoadjuvant therapy in women with stage II, III, or IV breast cancer.
* Correlate gene expression profiling of the primary breast cancer with axillary and sentinel lymph node status in these patients.

OUTLINE: This is a pilot study.

After neoadjuvant chemotherapy, patients undergo sentinel lymph node (SLN) mapping comprising technetium Tc 99m sulfur colloid injected into the subareolar area to identify the SLN. Within 1-2 hours after injection, patients undergo SLN biopsy followed immediately by definitive local surgery comprising modified radical mastectomy or breast segmentectomy with axillary lymph node dissection. SLN and axillary lymph nodes are examined by hematoxylin and eosin (H & E) staining for the presence or absence of metastases. If the lymph nodes are negative for tumor by H & E, the lymph nodes are further analyzed by immunohistochemistry. The primary tumor is analyzed by microarray analysis for gene expression profile determinations.

Patients are followed at 2-3 weeks after surgery.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma of the breast

  * Stage II, III, or IV infiltrating disease
  * Unilateral or bilateral AND unifocal or multifocal disease
* Received at least 1 course of prior preoperative therapy (chemotherapy, hormonal therapy, and/or biologic therapy) AND had any of the following responses:

  * Clinical complete response, partial response, no change, or disease progression
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 7.0 g/dL
* Platelet count > 50,000/mm^3
* WBC > 2,000/mm^3

Hepatic

* PT and PTT < 1.5 times normal

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* No prior definitive breast radiotherapy to the target breast

Surgery

* No prior axillary surgery on the side of the sentinel lymph node

Other

* More than 3 days since prior radionuclide scan (e.g., bone scan, positron-emission tomography scan, or MUGA scan)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N. Danforth, MD, MS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States